CLINICAL TRIAL: NCT04873388
Title: Biomarkers and Early Predictors of Prognostic Course, Response to Possible to Possible Treatments and Risk of Over-infection in Patients With COVID-19 Hospitalized in the Critical or Semi-intensive Area.
Brief Title: Early Predictors of Prognostic Course in Patients With COVID-19 in Critical or Semi-intensive Area.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-COVID-19
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Covid19; C-reactive Protein; Procalcitonin; D-dimer
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Results of the following assays will be retrieved for the different times of the study:
  * white blood cells (including data on leukocyte formula and lymphocyte subpopulations)
  * immunoglobulins
  * PCR, PCT, LDH, cardiac enzymes, NT-proBNP, ferritin
  * s-NA, s-K, blood glucose, renal function (creatinine, renal clearances, eGFR)
  * creatinine, renal clearance, eGFR
  * TSH, fT3, fT4
  * copeptin, MR-proADM The results of the laboratory data then, correlated with the parameters of cardiorespiratory function collected during the hospital stay and integrated with the prognostic scores of clinical use (Charlson, qSOFA, SOFA, SAPSII, APACHE, etc).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the recent literature is building a remarkable background to answer the many unknowns related to SARS-CoV-2 infection, it is absolutely necessary to finalize every clinical effort to collect data that may be useful, in a short time, to improve our knowledge of SARS-CoV-2 infection. Numerous biomarkers have been evaluated in the recent literature as being altered in patients with severe forms of COVID-19. Particularly, in the critical care area, the research of early predictors of mortality is essential for high-flow management of patients requiring invasive assisted ventilation and requiring invasive and non-invasive assisted ventilation, hemodynamic support, sometimes extracorporeal support (Extracorporeal Membrane Oxygenation, ECMO). The coordinated study of different biomarkers, in particular, if combined with each other, possibly even to constitute a possible score, could guide the correct allocation of patients between hospital departments and the appropriate management in intensive care units. appropriate management in intensive care units, as well as providing an early prognostic indication. prognostic indication. The combination of these biomarkers with routine clinical and laboratory data may further provide valuable information about their use in acute care and as progressive acute and as progressive monitoring over time.

Regarding the data of interest on the clinical trend, the evaluation of the respiratory support modalities, from the administration of oxygen therapy (by nasal cannulae or Venturi mask, or by high flow system - High Flow Nasal Cannula, HFNC), to CPAP support or by non-invasive or invasive ventilation, appears of particular importance.

Therefore, the present study will be conducted in sub-intensive as well as intensive care units, in order to evaluate different types of patients, and their possible evolution over time.

The comparison between the populations belonging to different areas of intensity of care will be able to describe the different populations. Data analysis will allow an evaluation of possible risk factors and prognostic determinants of the severity of the disease and its infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with clinical signs and symptoms of COVID-19, confirmed by nasopharyngeal swab RT-PCR of airways positive for SARS-CoV-2
* age > 18 years
* Hospitalization in the departments of the hospitals involved

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care areas (intensive care unit/intensive care unit) and semi-intensive care areas dedicated to the care of COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU inpatient mortality | 24 months
ICU inpatient length of stay | 24 months

SECONDARY OUTCOMES:
Incidence of over-infections (bacterial, viral, fungal), particularly of bacteremia and pneumonias associated with mechanical ventilation; observed infections' microbiological characteristics. | 24 months

OTHER OUTCOMES:
Identification of prognostic factors (biomarkers, clinical scores, respiratory support modalities, others). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Brazzi, Professor, Study Chair — University of Torino
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montrucchio G, Balzani E, Sales G, Bolla C, Sarda C, Della Selva A, Perotto M, Pomero F, Ravera E, Rumbolo F, Callegari T, Fanelli V, Mengozzi G, Brazzi L. Critical and non-critical coronavirus disease 2019 patients: which is the most predictive biomarker for disease severity and outcome?: A multicentre prospective cohort study comparing mid-regional pro-adrenomedullin, inflammatory and immunological patterns. Eur J Anaesthesiol Intensive Care. 2023 Nov 21;2(6):e0039. doi: 10.1097/EA9.0000000000000039. eCollection 2023 Dec. PMID 39916726